CLINICAL TRIAL: NCT01863615
Title: Bioequivalence Study for an Isotretinoin Pharmaceutical Preparation - Capsules. Crossover, Randomized, Single Dose, Two Treatments, Two Periods and Two Sequences With Meal (Breakfast) Study
Brief Title: Bioequivalence Study for an Isotretinoin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 116615
Record Dates: First submitted 2012-12-13; First posted 2013-05-29 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Skin Infections (Acne)
Keywords: pharmacokinetics; Isotretinoin; bioequivalence; Mexico
MeSH Terms: conditions — Cellulitis; Acne Vulgaris | interventions — Isotretinoin

ARMS (2):
- A(reference)/B(test) (Experimental): initial administration of reference and cross-over to test
  Interventions: Drug: Isotretinoin 40 mg
- B(test)/A(reference) (Experimental): initial administration of test and cross-over to reference
  Interventions: Drug: Isotretinoin 40 mg

INTERVENTIONS:
Drug: Isotretinoin 40 mg — Roaccutan 2 capsules of 20 mg; reference drug
  Other Names: Productos Roche; Roaccutan
Drug: Isotretinoin 40 mg — Oratane 2 capsules of 20 mg; test drug
  Other Names: Laboratorios Dermatologicos Darier SA de CV; Oratane

SUMMARY:
The objective of this study was to confirm if two formulations of isotretionin (capsules) are bioequivalent.

Test product was Oratane® 20 mg (Laboratorios Dermatológicos Darier) and reference product Roaccutan® 20 mg (Productos Roche). Two capsules administered together were the single dosage.

The study was prospective, open-label, randomized, crossover, single dose, with 02 treatments, 02 sequences and 02 periods, under fed conditions.

The population was composed of 36 healthy volunteers, male adults between 18-45 years.

The comparative bioavailability of the two formulations was evaluated based in statistical comparisons of relevant pharmacokinetic parameters, obtained from data of drug concentrations in blood.

ELIGIBILITY:
Inclusion Criteria:

Male volunteers. Ages between 18 and 45 years old. BMI (Body Mass Index) between 20 to 26 kg/m2. Anti-doping tests negative results. Clinical biochemical test values: Hematic Biometry, Urine Analysis, Biochemical Profile: (Glucose, Ureic Nitrogen, Urea, Creatinine, Uric Acid, Cholesterol, Triglycerides, Total Proteins, Albumin, Globulin, Bilirubin (total, indirect and direct), Alkaline Phosphatase, Lactic Dehydrogenase, AST, ALT, Calcium, Phosphorus, Sodium, Potassium, Chlorine and Iron), Ac VIH, AgsHB and RPR (luetic test), must fall within an interval between minimum and maximum values in connection to said tests accepted values.

Normal Electrocardiogram and Chest X-rays. In exception cases, accepted may be a candidate for which any previously mentioned test is exceeded regarding considered valid maximum and minimum accepted normal values, as long as it involves an isolated value and there are no other manifestations which could allow assuming that a given value is related to a disease or is remnant of another. These cases must be approved by clinical area and declared as "Non-clinically significant".

-

Exclusion Criteria:

Electrocardiographic Anomalies; radiological Anti-doping tests positive results, Positive results regarding RPR; VIH and AgsHB tests. Personal or family history of allergy to medication in question. Having any kind of allergy, since these persons are in higher risk of suffering from medicamentous allergy.

Tobacco use. Recreational drug use. Persons undergoing any medical treatment. Existence of concurrent or intercurrent disease. Existence of justified doubt regarding questionnaire answers truthfulness. Having participated in bioequivalence or bioavailability studies or having donated blood 2 months before the study.

Presence of clinically important gastrointestinal diseases or malabsorption history during the last year.

Presence of a medical condition requiring regular medication (with prescription or over-the- counter medication) with systemic absorption.

Narcotics or alcohol addiction history requiring treatment. Finally, excluded will be all those volunteers not meeting that established in Mexican Official Standard NOM-177-SSA1-1998.

-

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2011-08-26 (Actual); Primary Completion 2011-09-23 (Actual); Study Completion 2011-09-23 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (CMAX) of isotretinoin | 0.0, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36.0, 48.0, 60.0, 72.0 and 96.0 hours postdosage
  pharmacokinetics
Area under the plasma concentration versus time curve (AUC) of isotretionin | 0.0, 0.5, 1.0, 1.5, 2.0, 2.5, 3.0, 3.5, 4.0, 4.5, 5.0, 6.0, 7.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36.0, 48.0, 60.0, 72.0 and 96.0 hours postdosage
  pharmacokinetics

SECONDARY OUTCOMES:
Incidence od adverse events | 20 days
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Monterrey, Nuevo León, Mexico

REFERENCES:
- See also: Results for study 116615 can be found on the GSK Clinical Study Register. — https://www.gsk-clinicalstudyregister.com/study/116615?search=study&study_ids=116615#rs